CLINICAL TRIAL: NCT05508100
Title: A Phase 1, Open-Label, Multicenter Study Investigating Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IO-108 as Monotherapy and in Combination With Anti-PD-1 Monoclonal Antibody in Adult Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose Confirmation and Dose Expansion Phase 1 Study of IO-108 and IO-108 + Anti-PD-1 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune-Onc Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IO-108-CL-002
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A: IO-108 monotherapy dose confirmation (Experimental): Patients with advanced or metastatic solid tumors will be enrolled and treated with IO-108, intravenously, every 21 days.
  Interventions: Biological: IO-108
- Part B: IO-108 + anti-PD-1 dose confirmation. (Experimental): Patients will receive IO-108 in combination with with a fixed dose of pembrolizumab, intravenously, every 21 days; Patients will receive IO-108 in combination with with a fixed dose of tislelizumab, intravenously, every 21 days.
  Interventions: Biological: IO-108 + pembrolizumab; Biological: IO-108 + tislelizumab
- Part C: Dose expansion (Experimental): Patients with advanced or metastatic solid tumors who meet the specific criteria will be enrolled into one of the cohorts.
  Interventions: Biological: IO-108 + pembrolizumab; Biological: IO-108 + tislelizumab

INTERVENTIONS:
Biological: IO-108 — IO-108, intravenously, on Day 1 of each 21-day cycle.
  Arms: Part A: IO-108 monotherapy dose confirmation
Biological: IO-108 + pembrolizumab — IO-108, intravenously, on Day 1 of each 21-day cycle. Pembrolizumab will be administered intravenously on Day 1 of each 21-day cycle.
  Other Names: IO-108 + Keytruda®
  Arms: Part B: IO-108 + anti-PD-1 dose confirmation.; Part C: Dose expansion
Biological: IO-108 + tislelizumab — IO-108, intravenously, on Day 1 of each 21-day cycle. Tislelizumab will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Part B: IO-108 + anti-PD-1 dose confirmation.; Part C: Dose expansion

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, PK, and preliminary efficacy of IO-108 monotherapy and in combination with anti-PD-1 monoclonal antibody pembrolizumab or tislelizumab in adult patients with advanced solid tumors. The study will be conducted in 3 parts, including Part A IO-108 monotherapy dose confirmation; Part B IO-108 + anti-PD-1 dose confirmation, and Part C dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, and < 75.
2. Part A and Part B Cohort 1: Patients must have histologically or cytologically confirmed advanced or metastatic solid tumor and have failed, or have been intolerant for standard systemic therapy, or for whom no treatment known to confer clinical benefit exists.

   Part B Cohort 2 and Part C: Patient with advanced or metastatic solid tumor who meet the specific criteria.
3. Patients have at least 1 measurable disease per RECIST v1.1 as assessed by local clinical site.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
5. Patients must have adequate hematologic function, hepatic function and renal function.

Exclusion Criteria:

1. Patients who previously received a monoclonal antibody therapy targeting LILRB2/ILT4 (including IO-108).
2. Patients who received chemotherapy, radiotherapy, biologic therapy, targeted therapy, immunotherapy, or other investigational anti-cancer therapy < 4 weeks prior to their first day of study drug administration.
3. Requires systemic corticosteroids at a dose of >10 mg daily of prednisone or the dose equivalent to other systemic corticosteroid, or other immunosuppressive agents ≤ 14 days prior to the first dose.
4. History of radiation pneumonitis, non-infectious pneumonitis or interstitial lung disease expect for radioactive pulmonary fibrosis not requiring corticosteroid treatment.
5. Symptomatic central nervous system (CNS) metastases. Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) in patients treated with IO-108 | through study completion, an average of 2 years
  AE severity graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) in patients treated with IO-108 in combination with pembrolizumab or tislelizumab | through study completion, an average of 2 years
  AE severity graded by NCI CTCAE, Version 5.0
Preliminary anti-tumor activity of IO-108 in combination with pembrolizumab or tislelizumab | through study completion, an average of 2 years
  ORR is defined as the percentage of patients who have a complete response (CR) or a partial response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of IO-108 | through study completion, an average of 2 years
  Characterize the Cmax of IO-108 by successive sampling of blood at pre-specified time points
Steady state concentration of IO-108 | through study completion, an average of 2 years
  Characterize steady state concentration of IO-108 by successive sampling of blood at pre-specified time points
Anti-drug antibodies (ADA) of IO-108 | through study completion, an average of 2 years
  Determine the incidence and titer of ADAs against IO-108
Preliminary anti-tumor activity | through study completion, an average of 2 years
  Disease Control Rate, defined as the percentage of patients with CR, PR, or stable disease.
Preliminary anti-tumor activity | through study completion, an average of 2 years
  Progression-free Survival, defined as the time interval from the first dose date to the occurrence of disease progression or death of any cause

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - The First Affiliated Hospital of Fujian Medical University, Fujian, Fuzhou
  - 1st affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - 4th Hospitla of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Lin Yi Cancer Hospital, Linyi, Shandong
  - Shanghai Dong Fang Hospital, Shanghai, Shanghai Municipality
  - 1st Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Sir RUN RUN SHAW HOSPITAL, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No